CLINICAL TRIAL: NCT00345644
Title: A Non-invasive Evaluation of Bone Microarchitecture Modification in Osteopenic Postmenopausal Women by 3D Peripheral Quantitative Computed Tomography: A 24 Month, Monocenter Study Comparing Weekly Oral Risedronate 35 mg and Placebo
Brief Title: Risedronate in Osteopenic Postmenopausal Women
Acronym: OSMAUSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMR4003B_3507; EudraCT # :2005-005598-30
Record Dates: First submitted 2006-03-20; First posted 2006-06-28 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Osteoporosis
Keywords: Postmenopausal
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: risedronate
- 2 (Placebo Comparator)
  Interventions: Drug: risedronate placebo

INTERVENTIONS:
Drug: risedronate — risedronate sodium 35 mg tablets (once a week dose)
  Arms: 1
Drug: risedronate placebo — placebo for risedronate tablets (once a week dose)
  Arms: 2

SUMMARY:
The primary objective of this study is to compare risedronate 35 mg and placebo with respect to the percent change at 12 months for distal radius trabecular bone volume (BV/TV) in osteopenic postmenopausal women, as measured by three-dimensional peripheral quantitative computed tomography (3D pQCT).

The secondary objectives are to compare the percent change from Screening/Baseline between the 2 treatment groups for the following measurements:

* Bone mineral density of the lumbar spine, femoral neck, femoral trochanter, and total proximal femur using a dual energy X-ray absorptiometry (DXA) scan at 12 and 24 months;
* 3D pQCT analysis of distal radius and distal tibia bone microarchitecture data at 6, 12, and 24 months; and
* Bone turnover markers (BTMs) of:

  * fasting serum carboxyterminal cross linking telopeptide of type 1 bone collagen (CTX 1);
  * serum aminoterminal propeptide of type 1 procollagen (PINP); and
  * urine N-telopeptide cross-links (NTX) at 3, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Osteopenic, postmenopausal women, between 55 and 75 years of age with a body mass index (BMI) < 30 kg/m²

Exclusion Criteria:

* Clinical or radiological evidence of osteoporosis
* Severe renal impairment
* Serum 5-hydroxy vitamin D level < 15 ng/ml
* History of recent primary hyperparathyroidism or recent thyroid disorder
* History of any generalized bone disease
* Current use of glucocorticoids, estrogens, progestins, calcium supplements > 1 g/day, vitamin D supplements > 800 IU/day, parathyroid hormone (PTH), or any bisphosphonate for > 1 month at any time within the past 6 months.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Efficacy data : 3-D-pQCT Data-Microarchitectural Parameters (Distal Radius BV/TV Measurements) | BV/TV percent change from Baseline at distal radius as measured in the non dominant wrist at Month 12

SECONDARY OUTCOMES:
Tolerance data :collection of AEs, with special interest for upper gastrointestinal (UGI) AEs and clinical fractures | at all visits

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France